CLINICAL TRIAL: NCT06874127
Title: Establishment and Application of a Non-Invasive Dynamic Model for Fibrosis Regression in Patients with Chronic Hepatitis B
Brief Title: Non-Invasive Model for Fibrosis Regression in HBV Patients
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Sun Yameng, associate professor, Beijing Friendship Hospital
Other Study IDs: Z221100007422115; Z221100007422115 (Other Grant/Funding Number: Beijing Municipal Science & Technology Commission)
Record Dates: First submitted 2025-02-26; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Chronic Hepatitis B Virus (HBV) Infection; Liver Fibrosis
Keywords: chronic hepatitis B; Liver stiffness measurements; fibrosis regression; non-invasive
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Infections; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective cohort-derivation cohort
  Interventions: Drug: Nucleos(t)ide Analogs (NA)
- Retrospective cohort-validation cohort
  Interventions: Drug: Nucleos(t)ide Analogs (NA)

INTERVENTIONS:
Drug: Nucleos(t)ide Analogs (NA) — all patients received NAs

SUMMARY:
A total of 1000 chronic hepatitis B (CHB) patients with liver biopsy performed at least 1 year after antiviral therapy are retrospectively enrolled. All the patients received NAs treatment. Blood count, liver function test, alpha fetoprotein (AFP), prothrombin time, liver ultrasonography, liver stiffness measurement (LSM), Hepatitis B virus (HBV) DNA and HBV serological markers were collected. HBV-related endpoint events, including cirrhosis decompensations (ascites, esophageal variceal bleeding and hepatic encephalopathy), hepatocellular carcinoma (HCC), liver transplantation and liver-related death were collected. Fibrosis regression prediction model based on dynamic changes in liver stiffness will be developed based on the retrospective cohort. An independent cohort of CHB patients with liver biopsy performed at least 1 year after antiviral therapy will be retrospectively enrolled for model validation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver biopsy performed at least 1 year after antiviral therapy;
* Patients with liver biopsy or liver stiffness or aspartate aminotransferase (AST)-to-platelet (PLT) ratio index (APRI) before antiviral treatment.

Exclusion Criteria:

* Patients with decompensated cirrhosis (including ascites, hepatic encephalopathy, esophageal varices bleeding, hepatorenal syndrome, spontaneous bacterial peritonitis, or other complications of decompensated cirrhosis), hepatocellular carcinoma, or liver transplantation before liver biopsy;
* Patients with hepatitis C virus (HCV) or human immunodeficiency virus (HIV) infection, alcoholic liver disease, autoimmune liver disease, genetic liver disease, drug-induced liver injury, or other chronic liver diseases;
* Patients with malignant lesion on liver image;
* Patients with other uncured malignant tumors;
* Patients with severe heart, lung, kidney, brain, blood, neuropsychiatric or other organs diseases;
* Pregnant or lactating women;
* Patients with any other reasons not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CHB patients with liver biopsy performed at least 1 year after antiviral therapy
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of non-invasive model for fibrosis regression | 5 years
  Liver fibrosis regression was defined as decrease >= 1 point by Ishak fibrosis scoring system (range from 0 to 6, higher values represent a worse outcome) or Predominantly Regressive in P-I-R ( predominantly progressive, indeterminate and predominately regressive) score

SECONDARY OUTCOMES:
Incidence of HBV-related clinical endpoint events | 7 years
  clinical endpoint event includes: liver decompensations (ascites, esophageal variceal bleeding and hepatic encephalopathy), HCC, liver transplantation and liver-related death
Percentage of HBV-induced liver fibrosis regression | 5 years
  Liver fibrosis regression was defined as decrease >= 1 point by Ishak fibrosis scoring system (range from 0 to 6, higher values represent a worse outcome) or Predominantly Regressive in P-I-R ( predominantly progressive, indeterminate and predominately regressive) score
AUROC of non-invasive model for fibrosis regression | 5 years
  Liver fibrosis regression was defined as decrease >= 1 point by Ishak fibrosis scoring system (range from 0 to 6, higher values represent a worse outcome) or Predominantly Regressive in P-I-R ( predominantly progressive, indeterminate and predominately regressive) score
Sensitivity of non-invasive model for fibrosis regression | 5 years
  Liver fibrosis regression was defined as decrease >= 1 point by Ishak fibrosis scoring system (range from 0 to 6, higher values represent a worse outcome) or Predominantly Regressive in P-I-R ( predominantly progressive, indeterminate and predominately regressive) score
Specificity of non-invasive model for fibrosis regression | 5 years
  Liver fibrosis regression was defined as decrease >= 1 point by Ishak fibrosis scoring system (range from 0 to 6, higher values represent a worse outcome) or Predominantly Regressive in P-I-R ( predominantly progressive, indeterminate and predominately regressive) score

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No